CLINICAL TRIAL: NCT01416363
Title: A Single/Repeat Dose Study With Three Oral Formulations of Firategrast (Immediate Release Tablet, Modified Release Tablet, and Naso-gastric Infusion) in Healthy Male Volunteers
Brief Title: Healthy Volunteer Study Using 3 Different Formulations of Firategrast
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 115517
Record Dates: First submitted 2011-06-23; First posted 2011-08-15 (Estimated); Last update posted 2017-07-07 (Actual); Status verified 2017-07

CONDITIONS: Multiple Sclerosis, Relapsing-Remitting
Keywords: firategrast; pharmacokinetics, modified release, firategrast,; simulated gastro-retentive; pharmacokinetics; healthy volunteers, simulated gastro-retentive; healthy volunteers; modified release
MeSH Terms: conditions — Multiple Sclerosis, Relapsing-Remitting | interventions — Firategrast

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (9):
- Treatment Arm ACB: Part 1 (Experimental): Subjects will receive treatment sequence ACB; A : Firategrast immediate release tablet 1200 milligram (mg) once only orally, C : Firategrast simulated gastro-retentive solution 1200 mg once only by naso-gastric route, B : Firategrast 3 hour release tablet 1200 mg once only orally. There will be a washout period of 5 days between doses.
  Interventions: Drug: Firategrast immediate release tablet; Drug: Firategrast modified release tablet; Drug: Firategrast gastro-retentive solution
- Treatment Arm BAC: Part 1 (Experimental): Subjects will receive treatment sequence BAC; B : Firategrast 3 hour release tablet 1200 mg once only orally, A : Firategrast immediate release tablet 1200 mg once only orally, C : Firategrast simulated gastro-retentive solution 1200 mg once only by naso-gastric route. There will be a washout period of 5 days between doses.
  Interventions: Drug: Firategrast immediate release tablet; Drug: Firategrast modified release tablet; Drug: Firategrast gastro-retentive solution
- Treatment Arm CBA: Part 1 (Experimental): Subjects will receive treatment sequence CBA; C : Firategrast simulated gastro-retentive solution 1200 mg once only by naso-gastric route, B : Firategrast 3 hour release tablet 1200 mg once only orally, A : Firategrast immediate release tablet 1200 mg once only orally. There will be a washout period of 5 days between doses.
  Interventions: Drug: Firategrast immediate release tablet; Drug: Firategrast modified release tablet; Drug: Firategrast gastro-retentive solution
- Treatment Arm BCA: Part 1 (Experimental): Subjects will receive treatment sequence BCA; B : Firategrast 3 hour release tablet 1200 mg once only orally, C : Firategrast simulated gastro-retentive solution 1200 mg once only by naso-gastric route, A : Firategrast immediate release tablet 1200 mg once only orally. There will be a washout period of 5 days between doses.
  Interventions: Drug: Firategrast immediate release tablet; Drug: Firategrast modified release tablet; Drug: Firategrast gastro-retentive solution
- Treatment Arm CAB: Part 1 (Experimental): Subjects will receive treatment sequence CAB; C : Firategrast simulated gastro-retentive solution 1200 mg once only by naso-gastric route, A : Firategrast immediate release tablet 1200 mg once only orally, B : Firategrast 3 hour release tablet 1200 mg once only orally. There will be a washout period of 5 days between doses.
  Interventions: Drug: Firategrast immediate release tablet; Drug: Firategrast modified release tablet; Drug: Firategrast gastro-retentive solution
- Treatment Arm ABC: Part 1 (Experimental): Subjects will receive treatment sequence ABC; A : Firategrast immediate release tablet 1200 mg once only orally, B : Firategrast 3 hour release tablet 1200 mg once only orally, C : Firategrast simulated gastro-retentive solution 1200 mg once only by naso-gastric route. There will be a washout period of 5 days between doses.
  Interventions: Drug: Firategrast immediate release tablet; Drug: Firategrast modified release tablet; Drug: Firategrast gastro-retentive solution
- Treatment Arm D: Part 2 (Experimental): Subject will receive D: Firategrast immediate release tablet 600 mg twice daily for 7 days
  Interventions: Drug: Firategrast immediate release tablet; Drug: Firategrast modified release tablet; Drug: Firategrast gastro-retentive solution
- Treatment Arm E: Part 2 (Experimental): Subject will receive E: Firategrast 3 hour release tablet 1200 mg twice daily for 7 days
  Interventions: Drug: Firategrast immediate release tablet; Drug: Firategrast modified release tablet; Drug: Firategrast gastro-retentive solution
- Treatment Arm F: Part 2 (Experimental): Subject will receive F: Firategrast simulated gastro-retentive solution 1200 mg twice daily for 7 days
  Interventions: Drug: Firategrast immediate release tablet; Drug: Firategrast modified release tablet; Drug: Firategrast gastro-retentive solution

INTERVENTIONS:
Drug: Firategrast immediate release tablet — Firategrast immediate release tablet is white to pale cream colored 300 mg unit dose and subjects will administer it with 240 milliliter (mL) of water.
Drug: Firategrast modified release tablet — Firategrast modified release tablet is white to slightly colored 600 mg unit dose and subjects will administer it with 240 mL of water.
Drug: Firategrast gastro-retentive solution — Firategrast solution is clear colorless solution and subject will administer it via nasogastric route.

SUMMARY:
This study will investigate how 3 types of drug formulations are absorbed by the body. This study is termed 'open-label', which means volunteers will be aware of which treatment they are receiving. The study is split into 2 parts. Part 1, involves volunteers receiving 2 new formulations, as a single dose. There is no placebo (dummy-drug; no active ingredient) in this study. Volunteers will also receive a single dose of a formulation used in previous trials (reference formulation), so a proper comparison with the new formulations can be made. The new fomulations will be administered with food and the reference formulation will be given without food. In Part 2, volunteers will receive only one of the 3 formulations as a repeat dose for 7 days. Each of these doses will be given with food.

DETAILED DESCRIPTION:
The present study will be conducted in two parts in healthy male volunteers. Part 1 will investigate the pharmacokinetics and tolerability of single doses of firategrast administered as the existing immediate release tablet formulation, as a modified release tablet (3hr) formulation and as a simulated gastro-retentive formulation to be administered via a naso-gastric tube. Subjects will receive each formulation in a randomised 3-way single dose crossover fashion.

Part 2, based on the review of safety, tolerability and pharmacokinetic data from the first two study treatment periods of Part 1, will investigate the pharmacokinetics and tolerability of multiple doses of firategrast administered as the existing immediate release tablet formulation, as a modified release tablet (3hr) formulation and as simulated gastro-retentive formulation to be administered via naso-gastric tube for a period of 7 days.

ELIGIBILITY:
Inclusion Criteria:

* Male aged 18 to 65 yrs inclusive
* Healthy, as determined by study physician
* Capable of giving iformed consent

Exclusion Criteria:

* Positive drugs of abuse result
* Positive for HIV or Hepatitis B and/or C viruses
* History of alcohol consumption in excess of average recommended weekly intake (more than 12 units for males)
* Participation in a clinical trial within 30 days of scheduled first dose

Ages: 18 Years to 65 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2011-05-20 (Actual); Primary Completion 2011-09-17 (Actual); Study Completion 2011-09-17 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetic measures for single and repeat dose | Part 1: approx. 4 weeks, Part 2: approx 8 days
  Cmax of firategrast
PK measures for single and repeat dose | Part 1 approx 4 weeks, Part 2 approx 8 days
  AUC(0-t) of firategrast
Pharmacokinetic measurements for single and repeat dose | Part 1: approx 4 weeks, Part 2: approx 8 days
  AUC(0-24) of firategrast

SECONDARY OUTCOMES:
Safety & Tolerability in single and repeat doses | Part 1: approx. 4 weeks, Part 2: approx 8 days
  Adverse events, changes iin blood pressure, heart rate, ECGs, Haematology, clinical chemistry and urinalysis
CD34 positive cell count | Part 1 only approx 4 weeks
  as data permit - exploratory measure

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Randwick, New South Wales, Australia

REFERENCES:
- See also: Results for study 115517 can be found on the GSK Clinical Study Register. — https://www.gsk-clinicalstudyregister.com/study/115517?search=study&search_terms=115517#rs